CLINICAL TRIAL: NCT05349461
Title: Comparison of Post-operative Knee Range of Motion and Functions Between Intraoperative Complete and Incomplete Patellofemoral Articular Contacts in Patients Undergoing Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial
Brief Title: Comparison of Post-operative Knee Range of Motion and Functions Between Intraoperative Complete and Incomplete Patellofemoral Articular Contacts in Patients Undergoing Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA 010/2563
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-04

CONDITIONS: Complete Contact; Incomplete Contact

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete contact (Active Comparator)
  Interventions: Procedure: Complete patellofemoral articular contact
- Incomplete contact (Active Comparator)
  Interventions: Procedure: Incomplete patellofemoral articular contact

INTERVENTIONS:
Procedure: Complete patellofemoral articular contact — The patellofemoral condition is in constant contact with the femoral trochlea when the knee is bent from 30 to 90 degrees during the No thumb test.
  Arms: Complete contact
Procedure: Incomplete patellofemoral articular contact — The patellofemoral condition is in no constant contact with the femoral trochlea when the knee is bent from 30 to 90 degrees during the No thumb test.
  Arms: Incomplete contact

SUMMARY:
The purpose of this study is to compare clinical outcome in knee range of motion and functions between intraoperative complete and incomplete patellofemoral articular contacts

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty
* Age 50-80 year

Exclusion Criteria:

* Revision surgery
* Bilateral total knee arthroplasty
* History of patellar fracture
* History of patellar chondromalacia
* History of Patellar instability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Knee range of motion (ROM) | Change from baseline Knee range of motion (ROM) at 3 months, 6 months, and 12 months after surgery
  Goniometer measure range of motion (minimum 0, maximum 145)
Knee flexion | Change from baseline knee flexion at 3 months, 6 months, and 12 months after surgery
  Goniometer measure knee flexion (minimum 135, maximum 145)
Knee extension | Change from baseline knee extension at 3 months, 6 months, and 12 months after surgery
  Goniometer measure knee extension (minimum -10, maximum 0)

SECONDARY OUTCOMES:
Knee Society and Knee Society function score | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
New patellar score | Change from baseline new patellar score at 3 months, 6 months, and 12 months after surgery
  New patellar score (minimum 0, maximum 30)
Oxford knee score | Change from baseline Oxford knee score 3 months, 6 months, and 12 months after surgery
  Oxford knee score (minimum 0, maximum 48)
Prevalence of anterior knee pain ,AKP | Change from baseline Prevalence of anterior knee pain ,AKP 3 months, 6 months, and 12 months after surgery
  Prevalence of anterior knee pain ,AKP (minimum 0, maximum 10)

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — satitthh@hotmail.com
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand